CLINICAL TRIAL: NCT00558571
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of 4 Weeks Treatment With Three Oral Doses of BI 10773 as Tablets in Female and Male Patients With Type 2 Diabetes
Brief Title: 4 Week Treatment With Three Oral Doses of BI 10773 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1245.4; EudraCT No 2007-002685-36
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo to BI 10773
- BI 10773 low dose (Experimental)
  Interventions: Drug: BI 10773 low dose
- BI 10773 medium dose (Experimental)
  Interventions: Drug: BI 10773 medium dose
- BI 10773 high dose (Experimental)
  Interventions: Drug: BI 10773 high dose

INTERVENTIONS:
Drug: BI 10773 low dose
  Arms: BI 10773 low dose
Drug: placebo to BI 10773
  Arms: Placebo
Drug: BI 10773 medium dose
  Arms: BI 10773 medium dose
Drug: BI 10773 high dose
  Arms: BI 10773 high dose

SUMMARY:
Primary objective: safety and tolerability of BI 10773 in male and female patients with type 2 diabetes Secondary objective: pharmacokinetics and pharmacodynamics of BI 10773

ELIGIBILITY:
Inclusion Criteria:

* Male and postmenopausal or hysterectomised female patients with type 2 diabetes
* Age >18 and < 70 years
* BMI >18.5 and <40 kg/m2

Exclusion Criteria:

* Antidiabetic treatment with insulin or glitazones or with more than one oral hypoglycaemic agent;
* Fasted blood glucose > 240 mg/dl (>13.3 mmol/L) or a blood glucose level above 400 mg/dl (22.2 mmol/L) postprandially;
* HbA1c > 8.5 %

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Germany (3):
  - 1245.4.49003 Boehringer Ingelheim Investigational Site, Berlin
  - 1245.4.49002 Boehringer Ingelheim Investigational Site, Mainz
  - 1245.4.49001 Boehringer Ingelheim Investigational Site, Neuss

REFERENCES:
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Riggs MM, Staab A, Seman L, MacGregor TR, Bergsma TT, Gastonguay MR, Macha S. Population pharmacokinetics of empagliflozin, a sodium glucose cotransporter 2 inhibitor, in patients with type 2 diabetes. J Clin Pharmacol. 2013 Oct;53(10):1028-38. doi: 10.1002/jcph.147. Epub 2013 Aug 13. PMID 23940010

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo; 10mg Empagliflozin; 25mg Empagliflozin; 100mg Empagliflozin: Oral administration in the fasted state once daily
Period: Overall Study
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Started | 16 | 16 | 16 | 30
Completed | 16 | 16 | 16 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin | Total
Number analyzed (Participants) | 16 | 16 | 16 | 30 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (10.4) | 56.8 (8.7) | 56.1 (8.5) | 56.5 (8.2) | 56.7 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4 | 3 | 11
  Male | 15 | 13 | 12 | 27 | 67

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Drug Related Adverse Events
Description: number of subjects with investigator-defined drug-related adverse events.
Time Frame: from drug administration up to 6 weeks
Population: treated set: comprised all 78 patients who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
participants | 7 | 3 | 4 | 14

2. Primary Outcome: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinanalysis and ECG
Description: Clinical Relevant Abnormalities for Vital Signs, Blood Chemistry, Haematology, Urinanalysis and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: from drug administration up to 6 weeks
Population: treated set
Measure: Number; unit: participants
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
participants
  Lipase increased | 0 | 0 | 1 | 2
  Blood triglycerides increased | 0 | 1 | 0 | 0
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 1
  Ventricular extrasystoles | 0 | 1 | 0 | 0

3. Secondary Outcome: Cmax of Empagliflozin
Description: maximum concentration of the analyte in plasma after first dose (Cmax, Day 1 ) and at steady state over a uniform dosing interval (Cmax,ss, Day 28).
Time Frame: 0:05 before drug administration and 0:15 0:30 0:45 1:00 1:30 2:00 2:30 3:00 4:00 6:00 8:00 10:00 12:00 16:00 24:00 hours(h) after drug administration on day 1 and 28
Population: Pharmacokinetic (PK) analysis set: comprised all 62 patients who received Empagliflozin and had evaluable PK parameter data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 30
nmol/L
  Cmax | 309 (45.2) | 722 (20) | 2630 (25.8)
  Cmax,ss | 259 (24.8) | 687 (18.4) | 2390 (28.1)

4. Secondary Outcome: Tmax of Empagliflozin
Description: time from last dosing to maximum concentration of the analyte in plasma after first dose (Day 1), denoted by tmax; and at steady state (Day 28), denoted by tmax,ss.
Time Frame: 0:05 before drug administration and 0:15 0:30 0:45 1:00 1:30 2:00 2:30 3:00 4:00 6:00 8:00 10:00 12:00 16:00 24:00 h after drug administration on day 1 and 28
Population: PK analysis set
Measure: Median (Full Range); unit: hours
Arm/Group | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 30
hours
  tmax | 1.50 (29.8) [1.00 to 2.50] | 1.50 (28.7) [0.75 to 2.00] | 1.50 (30.9) [0.75 to 3.00]
  tmax,ss | 1.50 (13) [0.98 to 4.00] | 1.50 (14.9) [0.75 to 3.02] | 1.50 (18.7) [0.75 to 6.00]

5. Secondary Outcome: t1/2 of Empagliflozin
Description: terminal half-life of the analyte in plasma after first dose (Day 1), denoted by t1/2; and at steady state (Day 28), denoted by t1/2,ss.
Time Frame: as for outcome 4
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 30
hours
  t1/2 | 8.69 (12.90) | 8.16 (14.50) | 8.53 (18.50)
  t1/2,ss | 12.20 (41.40) | 12.70 (32.70) | 15.00 (44.30)

6. Secondary Outcome: AUC0-∞ of Empagliflozin
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) and over a uniform dosing interval τ at steady state (AUCτ,ss)
Time Frame: 0:05 before drug administration and 0:15 0:30 0:45 1:00 1:30 2:00 2:30 3:00 4:00 6:00 8:00 10:00 12:00 16:00 24:00 h after drug administration on day 1
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 30
nmol*h/L
  AUC0-∞ | 1740 (16.4) | 4340 (23.1) | 18000 (24.3)
  AUCτ,ss | 1870 (15.9) | 4740 (21.2) | 18700 (25.2)

7. Secondary Outcome: CL/F of Empaglifozin
Description: apparent clearance of the analyte in plasma after first dose (CL/F) and at steady state (CL/F,ss)
Time Frame: as for outcome 4
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 30
mL/min
  CL/F | 218 (15.3) | 223 (21.2) | 215 (20.8)
  CL/F,ss | 202 (15.9) | 203 (21.4) | 208 (22)

8. Secondary Outcome: fe0-24 of Empagliflozin
Description: Fraction of analyte eliminated in urine from time point 0 to 24h after first dose (fe0-24) and at steady state (fe0-24,ss)
Time Frame: as for outcome 4
Population: PK analysis set for patients who have fe data at day 1 and day 28
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of Empagliflozin
Arm/Group | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 15 | 16 | 30
percentage of Empagliflozin
  fe0-24 (N=14,16,30) | 12.5 (24) | 13.3 (24.5) | 13.7 (34.1)
  fe0-24,ss | 18.3 (25) | 17.8 (17.8) | 17.5 (28.3)

9. Secondary Outcome: LI (Linearity Index).
Description: The linearity index is defined as AUC0-τ divided by AUC0-∞ both at steady state.
Time Frame: 0:05 before drug administration and 0:15 0:30 0:45 1:00 1:30 2:00 2:30 3:00 4:00 6:00 8:00 10:00 12:00 16:00 after drug administration on day 1 and 28
Population: PK analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 30
ratio | 1.09 (11.1) | 1.1 (12.5) | 1.04 (9.21)

10. Secondary Outcome: Ae0-24 of Glucose
Description: Amount of glucose eliminated in urine over the time interval 0 to 24h on day -2, -1, 1, 27 and 28. (Urinary Glucose Excretion)
Time Frame: Day -2 and 27: -2 to 0, 0 to 5, 5 to 12 and 12 to 24h; Day -1 and 1: 0 to 5, 5 to 12 and 12 to 24; Day 28: 0 to 5, 5 to 12, 12 to 24, 24 to 36, 36 to 48 and 48 to 72h
Population: PD analysis set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
mg
  Ae0-24 on day -2 (N=15,16,15,26) | 4270 (185) | 7760 (161) | 5340 (123) | 6050 (190)
  Ae0-24 on day -1 (N=13,15,16,25) | 6490 (136) | 8450 (114) | 8150 (91) | 6190 (134)
  Ae0-24 on day 1 (N=15,15,16,29) | 3970 (197) | 81500 (35.7) | 95700 (30.4) | 87000 (36.9)
  Ae0-24 on day 27 (N=14,13,14,27) | 3790 (296) | 78000 (44.1) | 82900 (32.9) | 81300 (50.1)
  Ae0-24 on day 28 (N=13,13,11,23) | 6310 (230) | 75400 (44.6) | 83400 (26.4) | 73900 (61.6)

11. Secondary Outcome: Fasting Plasma Glucose (FPG)
Description: fasting plasma glucose on day -1 (baseline) and change from baseline to day 28
Time Frame: in the morning of days -1 and 28
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 29
mg/dL
  baseline (day -1) | 153.87 (40.53) | 186.18 (92.96) | 167.49 (39.61) | 149.92 (31.65)
  change from baseline to day 28 (N=15, 15, 16, 28) | -4.08 (27.08) | -43.7 (81.81) | -34.22 (26.44) | -28.69 (18.25)

12. Secondary Outcome: Mean Daily Glucose (MDG) Measured in Blood
Description: change from baseline in MDG on the days 1, 7, 14, 21 and 27. Baseline is defined as day -2.
Time Frame: 0:00, 2:30, 5:00, 7:00, 10:00, 12:00, 13:30, 24:00 h after drug administration on day -2. 0:05 h before drug administration and 2:30, 5:00, 7:00, 10:00, 12:00, 13:30, 24:00 h after drug administration on day 1, 7, 14, 21 and 27
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
mg/dL
  baseline (day -2) | 152.06 (41.49) | 164.83 (43.18) | 166.26 (35.86) | 149.43 (34.94)
  change from baseline to day 1 | 2.13 (18.37) | -14.69 (15.81) | -23.51 (17.26) | -23.02 (16.72)
  change from baseline to day 7 | -2.4 (15.78) | -25.45 (23.2) | -28.58 (17.6) | -21.17 (21.95)
  change from baseline to day 14 | 2.68 (28.05) | -26.97 (27.9) | -20.43 (24.69) | -12.03 (28.51)
  change from baseline to day 21 | -3.41 (30.46) | -26.47 (31.71) | -19.68 (24.94) | -13.93 (24.46)
  change from baseline to day 27 | -4.69 (32.01) | -19.57 (28) | -26.37 (18.74) | -23.87 (18.44)

13. Secondary Outcome: Insulin AUEC0-5
Description: change in AUEC0-5 from baseline on day 28. Baseline is defined as day -1.
Time Frame: 0:00, 2:30, 5:00, 7:00, 10:00, 12:00 after drug administration on day -1. 0:05 before drug administration and 2:30, 5:00, 7:00, 10:00, 12:00 after drug administration on day 28.
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: µU*h/mL
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
µU*h/mL
  baseline (day -1) | 108.16 (70.85) | 117.34 (54.36) | 102.44 (65.8) | 121.53 (101.07)
  change from baseline to day 28 (N=16, 16, 16, 29) | 24.37 (99.44) | 3.24 (91.07) | 3.8 (73.66) | 8.83 (67.79)

14. Secondary Outcome: Insulin Emax (Maximum Measured Effect)
Description: change in Emax from baseline on day 28. Baseline is defined as day -1
Time Frame: as for outcome 13
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
µU/mL
  baseline (day -1) | 50.78 (28.35) | 48.09 (23.38) | 46.13 (24.7) | 53.06 (43.3)
  change from baseline to day 28 (N=16, 16, 16, 29) | 7.77 (30.73) | 0.55 (36.94) | -0.46 (28.46) | 2.92 (32.52)

15. Secondary Outcome: Fasting Insulin
Description: Change from baseline to the days 1, 7, 14, 21 and 28. Baseline is defined as day -1.
Time Frame: in the morning of days -1( baseline), 1, 7, 14, 21 and 28
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: µU/mL
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
µU/mL
  baseline (day -1) (N=12,12,14,23) | 10 (4.37) | 11.43 (6.23) | 8.74 (4.13) | 9.3 (5.14)
  change from baseline to day 1 (N=11,12,14,22) | -1.08 (2.9) | -1.56 (3.97) | -1.1 (2.29) | 0.15 (4.51)
  change from baseline to day 7 (N=9,10,9,18) | 0.48 (2.56) | -2.49 (6.01) | -1 (3.36) | -0.2 (6.58)
  change from baseline to day 14 (N=12,11,14,22) | 2.32 (4.68) | -1.16 (4.58) | 0.18 (2.74) | 1.37 (4.75)
  change from baseline to day 21 (N=10,11,14,21) | 1.84 (4.76) | -0.17 (6.35) | -1.21 (2.85) | 1.53 (5.87)
  change from baseline to day 28 (N=11,11,12,20) | -1.2 (1.74) | -2.89 (4.68) | -1.73 (3.64) | -2.1 (4.46)

16. Secondary Outcome: Glucagon Emax (Maximum Measured Effect)
Description: Change from baseline (day -1) in Emax on day 28.
Time Frame: 0:00, 2:30, 5:00, 7:00, 10:00, 12:00, 24:00 h after drug administration on day -1. 0:05 before drug administration and 2:30, 5:00, 7:00, 10:00, 12:00 after drug administration on day 28.
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
ng/L
  baseline (day -1) | 80.35 (18.01) | 90.58 (19.63) | 82.75 (17.79) | 86.98 (22.51)
  change from baseline to day 28 (N=14, 14, 16, 28) | 12.44 (28.69) | 13.69 (23.96) | 7.84 (16.66) | 6.84 (21.45)

17. Secondary Outcome: Glucagon AUEC0-5
Description: Change from baseline (day -1) in AUEC0-5 on day 28.
Time Frame: as for outcome 13
Population: Pharmacodynamic (PD) analysis set: All patients who receive at least one dose of study medication (active drug or placebo) and had some PD data were included in the pharmacodynamic analysis.
Measure: Mean (Standard Deviation); unit: ng*h/L
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
ng*h/L
  baseline (day -1) | 290.66 (74.99) | 310.76 (72.1) | 291.09 (104.11) | 303.06 (75.4)
  change from baseline to day 28 (N=14, 14, 16, 28) | 9.01 (81.1) | 59.69 (89.52) | 33.6 (73.09) | 40.65 (75.72)

18. Secondary Outcome: Fructosamine
Description: change from baseline to days 14 and 18. Baseline is defined as day -1.
Time Frame: day -1 (baseline), 14 and 28
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 16 | 16 | 30
µmol/L
  baseline (day -1) | 237.27 (33.97) | 251.88 (39.19) | 257.88 (53.64) | 237.07 (41.48)
  change from baseline to day 14 (N=14, 16, 15, 29) | 19.57 (24.67) | 24.75 (21.55) | 13.07 (20.83) | 18.31 (22)
  change from baseline to day 28 (N=14, 15, 16, 28) | -23.57 (28.67) | -24.33 (29.98) | -22.06 (32.89) | -26.29 (31.04)

19. Secondary Outcome: HbA1c
Description: change from baseline on day 28. Baseline is defined as day -1.
Time Frame: in the morning of days -1 and 28
Population: PD analysis set
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Number analyzed (Participants) | 16 | 15 | 16 | 30
percentage of hemoglobin
  baseline (day -1) | 6.89 (0.91) | 7.15 (0.67) | 7.45 (0.8) | 7.1 (0.88)
  change from baseline to day 28 (N=13, 13, 15, 28) | -0.18 (0.62) | -0.27 (0.36) | -0.22 (0.32) | -0.36 (0.31)

ADVERSE EVENTS:
Time Frame: From screening (35 to 15 days before treatment administration) until the end of study examination (35 to 41 days after treatment administration)
Description: Patients were required to report spontaneously any AEs, including the time of onset, duration and intensity of these events. Each patient could be assessed by the investigator whenever necessary.
Arm/Group | Placebo | 10mg Empagliflozin | 25mg Empagliflozin | 100mg Empagliflozin
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/30
Other Adverse Events (participants affected / at risk) | 10/16 | 8/16 | 9/16 | 18/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | 10mg Empagliflozin (N=16) | 25mg Empagliflozin (N=16) | 100mg Empagliflozin (N=30)
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Fatigue (General disorders) | 1 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 2 | 2 | 3
Polyuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Balanitis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.